CLINICAL TRIAL: NCT06130397
Title: FRACT-AI: Evaluating the Impact of Artificial Intelligence-Enhanced Image Analysis on the Diagnostic Accuracy of Frontline Clinicians in the Detection of Fractures on Plain X-Ray
Brief Title: AI Assisted Detection of Fractures on X-Rays (FRACT-AI)
Acronym: FRACT-AI
Status: Completed | Type: Observational
Sponsor: Oxford University Hospitals NHS Trust (Other)
Collaborators: Gleamer (Industry)
Responsible Party: Principal Investigator, Alex Novak, Primary Investigator, Oxford University Hospitals NHS Trust
Other Study IDs: 310995-C
Record Dates: First submitted 2023-11-08; First posted 2023-11-14 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Fracture; Bone Fracture; Dislocation; Fracture Multiple; Fractures, Closed; Fractures, Open
Keywords: radiology; emergency medicine; artificial intelligence; XRays; Fractures
MeSH Terms: conditions — Fractures, Bone; Joint Dislocations; Fractures, Multiple; Fractures, Closed; Fractures, Open

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Readers/participants: Reader Selection: 18 readers will be selected from the following five clinical specialty groups (3 readers each):
  * Emergency Medicine
  * Trauma and Orthopaedic Surgery
  * Emergency Nurse Practitioners
  * Physiotherapy
  * General Radiology
  * Radiographers
  And from the following level of seniority/experience:
  * Consultant/Senior/Equivalent - >10yrs experience
  * Middle Grade/Registrar/Equivalent - 5-10yrs experience
  * Junior Grade/Senior House Officer/Equivalent - <5yrs experience
  Each specialty reader group will include 1 reader at each level of experience.
  Readers will be recruited from across 5 NHS organisations which comprise the Thames Valley Emergency Medicine Research Network (www.TaVERNresearch.org):
  * Oxford University Hospitals NHS Foundation Trust
  * Royal Berkshire NHS Foundation Trust
  * Buckinghamshire Healthcare NHS Trust
  * Frimley Health NHS Foundation Trust
  * Milton Keynes University Hospital NHS Foundation Trust
  Interventions: Other: Cases reading
- Ground truthers: Two consultant musculoskeletal radiologists. A third senior musculoskeletal radiologist's opinion (>20 years experience) will undertake arbitration.
  Interventions: Other: Ground truthing

INTERVENTIONS:
Other: Cases reading — The reading will be done remotely via the Report and Image Quality Control site (www.RAIQC.com), an online platform allowing medical imaging viewing and reporting. Participants can work from any location, but the work must be done from a computer with internet access. For avoidance of doubt, the work cannot be performed from a phone or tablet.
  The project is divided into two phases and participants are required to complete both phases. The estimated total involvement in the project is up to 20-24 hours.
  Phase 1: Time allowed: 2 weeks
  - Participants must review 500 X-rays and express a clinical opinion through a structured reporting template (multiple choice, no open text required).
  Rest/washout period - Time allowed: 4 weeks, to mitigate the effects of recall bias.
  Phase 2 - Time allowed: 2 weeks
  - Review 500 X-rays together with an AI report for each case and express their clinical opinion through the same structured reporting template used in Phase 1.
  Groups: Readers/participants
Other: Ground truthing — Two consultant musculoskeletal radiologists will independently review the images to establish the 'ground truth' findings on the XRs, where a consensus is reached this will then be used as the reference standard. In the case of disagreement, a third senior musculoskeletal radiologist's opinion (>20 years experience) will undertake arbitration. A difficulty score will be assigned to each abnormality by the ground truthers using a 4-point Likert scale (1 being easy/obvious to 4 being hard/poorly visualised).
  Groups: Ground truthers

SUMMARY:
This study has been added as a sub study to the Simulation Training for Emergency Department Imaging 2 study (ClinicalTrials.gov ID NCT05427838). This work aims to evaluate the impact of an Artificial Intelligence (AI)-enhanced algorithm called Boneview on the diagnostic accuracy of clinicians in the detection of fractures on plain XR (X-Ray). The study will create a dataset of 500 plain X-Rays involving standard images of all bones other than the skull and cervical spine, with 50% normal cases and 50% containing fractures. A reference 'ground truth' for each image to confirm the presence or absence of a fracture will be established by a senior radiologist panel. This dataset will then be inferenced by the Gleamer Boneview algorithm to identify fractures. Performance of the algorithm will be compared against the reference standard. The study will then undertake a Multiple-Reader Multiple-Case study in which clinicians interpret all images without AI and then subsequently with access to the output of the AI algorithm. 18 clinicians will be recruited as readers with 3 from each of six distinct clinical groups: Emergency Medicine, Trauma and Orthopedic Surgery, Emergency Nurse Practitioners, Physiotherapy, Radiology and Radiographers, with three levels of seniority in each group. Changes in reporting accuracy (sensitivity, specificity), confidence, and speed of readers in two sessions will be compared. The results will be analyzed in a pooled analysis for all readers as well as for the following subgroups: Clinical role, Level of seniority, Pathological finding, Difficulty of image. The study will demonstrate the impact of an AI interpretation as compared with interpretation by clinicians, and as compared with clinicians using the AI as an adjunct to their interpretation. The study will represent a range of professional backgrounds and levels of experience among the clinical element. The study will use plain film x-rays that will represent a range of anatomical views and pathological presentations, however x-rays will present equal numbers of pathological and non-pathological x-rays, giving equal weight to assessment of specificity and sensitivity. Ethics approval has already been granted, and the study will be disseminated through publication in peer-reviewed journals and presentation at relevant conferences.

ELIGIBILITY:
Inclusion Criteria:

* Emergency medicine doctors, trauma and orthopaedic surgeons, emergency nurse practitioners, physiotherapists, general radiologists and radiographers reviewing X-rays as part of their routine clinical practice.
* Currently working in the National Health Service (NHS).

Exclusion Criteria:

* Non-radiology physicians with previous formal postgraduate XR reporting training.
* Non-radiology physicians with previous career in radiology

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Emergency medicine doctors, trauma and orthopaedic surgeons, emergency nurse practitioners, physiotherapists, general radiologists and radiographers reviewing X-rays as part of their routine clinical practice, currently working in the National Health Service (NHS).
  Readers will be recruited from across 5 NHS organisations which comprise the Thames Valley Emergency Medicine Research Network (www.TaVERNresearch.org):
  * Oxford University Hospitals NHS Foundation Trust
  * Royal Berkshire NHS Foundation Trust
  * Buckinghamshire Healthcare NHS Trust
  * Frimley Health NHS Foundation Trust
  * Milton Keynes University Hospital NHS Foundation Trust
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2024-02-08 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
Performance of AI algorithm: sensitivity | During 4 weeks of reading time
  Evaluation of the Gleamer Boneview algorithm will be performed comparing it to the reference standard in order to determine sensitivity.
Performance of AI algorithm: specificity | During 4 weeks of reading time
  Evaluation of the Gleamer Boneview will be performed comparing it to the reference standard in order to determine specificity.
Performance of AI algorithm: Area under the ROC Curve (AU ROC) | During 4 weeks of reading time
  Evaluation of the Gleamer Boneview algorithm will be performed comparing it to the reference standard. Continuous probability score from the algorithm will be utilised for the ROC analyses, while binary classification results with a predefined operating cut-off will be used for evaluation of sensitivity, specificity, positive predictive value, and negative predictive value.
Performance of readers with and without AI assistance: Sensitivity | During 4 weeks of reading time
  The study will include two sessions (with and without AI overlay), with all 18 readers reviewing all 500 XR cases each time separated by a washout period to mitigate recall bias. The cases will be randomised between the two reads and for every reader.
Performance of readers with and without AI assistance: Specificity | During 4 weeks of reading time
  The study will include two sessions (with and without AI overlay), with all 18 readers reviewing all 500 XR cases each time separated by a washout period to mitigate recall bias. The cases will be randomised between the two reads and for every reader.
Performance of readers with and without AI assistance: Area under the ROC Curve (AU ROC) | During 4 weeks of reading time
  The study will include two sessions (with and without AI overlay), with all 18 readers reviewing all 500 XR cases each time separated by a washout period to mitigate recall bias. The cases will be randomised between the two reads and for every reader.
Reader speed with vs without AI assistance. | During 4 weeks of reading time
  Mean time taken to review a XR, with vs without AI assistance.

CONTACTS AND LOCATIONS:
Locations (1):
- Oxford University Hospitals NHS Foundation Trust, Oxford, Oxfordshire, United Kingdom

REFERENCES:
- [Background] Hussain F, Cooper A, Carson-Stevens A, Donaldson L, Hibbert P, Hughes T, Edwards A. Diagnostic error in the emergency department: learning from national patient safety incident report analysis. BMC Emerg Med. 2019 Dec 4;19(1):77. doi: 10.1186/s12873-019-0289-3. PMID 31801474
- [Background] Donaldson LJ, Reckless IP, Scholes S, Mindell JS, Shelton NJ. The epidemiology of fractures in England. J Epidemiol Community Health. 2008 Feb;62(2):174-80. doi: 10.1136/jech.2006.056622. PMID 18192607
- [Background] National Clinical Guideline Centre (UK). Fractures (Non-Complex): Assessment and Management. London: National Institute for Health and Care Excellence (NICE); 2016 Feb. Available from http://www.ncbi.nlm.nih.gov/books/NBK344251/ PMID 26913322
- [Background] Blazar E, Mitchell D, Townzen JD. Radiology Training in Emergency Medicine Residency as a Predictor of Confidence in an Attending. Cureus. 2020 Jan 9;12(1):e6615. doi: 10.7759/cureus.6615. PMID 32064195
- [Background] Snaith B, Hardy M. Emergency department image interpretation accuracy: The influence of immediate reporting by radiology. Int Emerg Nurs. 2014 Apr;22(2):63-8. doi: 10.1016/j.ienj.2013.04.004. Epub 2013 May 30. PMID 23726985
- [Background] York TJ, Jenkins PJ, Ireland AJ. Reporting Discrepancy Resolved by Findings and Time in 2947 Emergency Department Ankle X-rays. Skeletal Radiol. 2020 Apr;49(4):601-611. doi: 10.1007/s00256-019-03317-7. Epub 2019 Nov 21. PMID 31754742
- [Background] van Leeuwen KG, Schalekamp S, Rutten MJCM, van Ginneken B, de Rooij M. Artificial intelligence in radiology: 100 commercially available products and their scientific evidence. Eur Radiol. 2021 Jun;31(6):3797-3804. doi: 10.1007/s00330-021-07892-z. Epub 2021 Apr 15. PMID 33856519
- [Background] Duron L, Ducarouge A, Gillibert A, Laine J, Allouche C, Cherel N, Zhang Z, Nitche N, Lacave E, Pourchot A, Felter A, Lassalle L, Regnard NE, Feydy A. Assessment of an AI Aid in Detection of Adult Appendicular Skeletal Fractures by Emergency Physicians and Radiologists: A Multicenter Cross-sectional Diagnostic Study. Radiology. 2021 Jul;300(1):120-129. doi: 10.1148/radiol.2021203886. Epub 2021 May 4. PMID 33944629
- [Background] Fenton JJ, Taplin SH, Carney PA, Abraham L, Sickles EA, D'Orsi C, Berns EA, Cutter G, Hendrick RE, Barlow WE, Elmore JG. Influence of computer-aided detection on performance of screening mammography. N Engl J Med. 2007 Apr 5;356(14):1399-409. doi: 10.1056/NEJMoa066099. PMID 17409321
- [Background] Chilamkurthy S, Ghosh R, Tanamala S, Biviji M, Campeau NG, Venugopal VK, Mahajan V, Rao P, Warier P. Deep learning algorithms for detection of critical findings in head CT scans: a retrospective study. Lancet. 2018 Dec 1;392(10162):2388-2396. doi: 10.1016/S0140-6736(18)31645-3. Epub 2018 Oct 11. PMID 30318264
- [Background] Patel MR, Norgaard BL, Fairbairn TA, Nieman K, Akasaka T, Berman DS, Raff GL, Hurwitz Koweek LM, Pontone G, Kawasaki T, Sand NPR, Jensen JM, Amano T, Poon M, Ovrehus KA, Sonck J, Rabbat MG, Mullen S, De Bruyne B, Rogers C, Matsuo H, Bax JJ, Leipsic J. 1-Year Impact on Medical Practice and Clinical Outcomes of FFRCT: The ADVANCE Registry. JACC Cardiovasc Imaging. 2020 Jan;13(1 Pt 1):97-105. doi: 10.1016/j.jcmg.2019.03.003. Epub 2019 Mar 17. PMID 31005540
- [Background] Obuchowski NA, Bullen J. Multireader Diagnostic Accuracy Imaging Studies: Fundamentals of Design and Analysis. Radiology. 2022 Apr;303(1):26-34. doi: 10.1148/radiol.211593. Epub 2022 Feb 15. PMID 35166584
- [Background] Smith BJ, Hillis SL. Multi-reader multi-case analysis of variance software for diagnostic performance comparison of imaging modalities. Proc SPIE Int Soc Opt Eng. 2020 Feb;11316:113160K. doi: 10.1117/12.2549075. Epub 2020 Mar 16. PMID 32351258
- [Derived] Novak A, Hollowday M, Espinosa Morgado AT, Oke J, Shelmerdine S, Woznitza N, Metcalfe D, Costa ML, Wilson S, Kiam JS, Vaz J, Limphaibool N, Ventre J, Jones D, Greenhalgh L, Gleeson F, Welch N, Mistry A, Devic N, Teh J, Ather S. Evaluating the impact of artificial intelligence-assisted image analysis on the diagnostic accuracy of front-line clinicians in detecting fractures on plain X-rays (FRACT-AI): protocol for a prospective observational study. BMJ Open. 2024 Sep 5;14(9):e086061. doi: 10.1136/bmjopen-2024-086061. PMID 39237277
- See also: 3. Clinical negligence claims in Emergency Departments in England. Report 2 of 3: Missed fractures. NHS Resolution. March 2022 — https://resolution.nhs.uk/wp-content/uploads/2022/03/2-NHS-Resolution-ED-report-Missed-Fractures.pdf
- See also: 11. The NICE Evidence Standards Framework for digital health and care technologies. (ECD7) Last Updated: 9 August — http://www.nice.org.uk/corporate/ecd7